CLINICAL TRIAL: NCT03693612
Title: A Phase I/II, Open-label, Two Part Study of GSK3359609 in Combination With Tremelimumab in Participants With Selected, Advanced Solid Tumors
Brief Title: GSK3359609 Plus Tremelimumab for the Treatment of Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207871
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms
Keywords: advanced solid tumor; Head and Neck Squamous Cell Carcinoma; standard of care; GSK3359609; urothelial carcinoma of the upper and lower urinary tract; non-small cell lung cancer; cutaneous melanoma; Tremelimumab; clear cell renal carcinoma; castrate resistant prostate adenocarcinoma
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell | interventions — tremelimumab; Docetaxel; Paclitaxel; Cetuximab

STUDY DESIGN:
Intervention Model Description: In Part 1, dose escalation will occur using a zone based approach. Part 2 will be randomized, parallel group study wherein the subjects will be randomized in a ratio of 2:1 to either recommended Phase 2 dose combination of GSK3359609 and tremelimumab or SOC (paclitaxel, docetaxel or cetuximab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: feladilimab +tremelimumab (Experimental): In Part 1, subjects with advanced selected solid tumors will be enrolled. Subjects will be administered escalating doses of feladilimab and tremelimumab in combination. feladilimab will be administered every 3 weeks and tremelimumab will be administered every 3 weeks for 6 doses and every 12 weeks thereafter.
  Interventions: Drug: feladilimab; Drug: Tremelimumab
- Part 2: feladilimab +tremelimumab (Experimental): In Part 2, subjects with R/R HNSCC who have disease progression after receiving at least one platinum-based chemotherapy and at least one anti-PD-1/PD-L1 will be enrolled. Subjects will be administered feladilimab in combination with tremelimumab at recommended Phase 2 dose as determined from Part 1.
  Interventions: Drug: feladilimab; Drug: Tremelimumab
- Part 2: SOC (Active Comparator): In Part 2, subjects with R/R HNSCC who have disease progression after receiving at least one platinum-based chemotherapy and at least one anti-PD-1/PD-L1 will be enrolled. Subjects will be administered a single agent SOC therapy of either paclitaxel, docetaxel or cetuximab as per the investigators choice.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Cetuximab

INTERVENTIONS:
Drug: feladilimab — feladilimab is humanized anti-ICOS agonist immunoglobulin G (IgG) 4 monoclonal antibody (mAb), which will be administered as an intravenous (IV) infusion once every 3 weeks.
  Arms: Part 1: feladilimab +tremelimumab; Part 2: feladilimab +tremelimumab
Drug: Tremelimumab — Tremelimumab is humanized anti-CTLA-4 IgG2 mAb, which will be administered as an IV infusion once every 3 weeks for 6 doses, thereafter once every 12 weeks .
  Arms: Part 1: feladilimab +tremelimumab; Part 2: feladilimab +tremelimumab
Drug: Docetaxel — Docetaxel is a microtubule stabilizer which will be administered as an IV infusion once every 3 weeks at a dose of 75 milligrams per meter square (mg/m^2).
  Arms: Part 2: SOC
Drug: Paclitaxel — Paclitaxel is a microtubule stabilizer which will be administered as an IV infusion once weekly at a dose of 80 mg/m^2.
  Arms: Part 2: SOC
Drug: Cetuximab — Cetuximab is a recombinant, human/mouse chimeric anti-estimated glomerular filtration rate (EGFR) mAb. Cetuximab will be administered at a loading dose of 400 mg/m^2 followed by 250 mg/m^2 once weekly.
  Arms: Part 2: SOC

SUMMARY:
The purpose of this study is to evaluate if the combination of GSK3359609 and tremelimumab is safe and tolerable (Part 1) and provides significant survival benefit to subjects with relapsed/refractory (R/R) Head and Neck Squamous Cell Carcinomas (HNSCC) to warrant further clinical investigation (Part 2). Part 1 (dose escalation) will enroll subjects with advanced, selected solid tumors. Subjects will receive escalating doses of GSK3359609 and tremelimumab in combination in Part 1. Part 2 is randomized expansion and will enroll subjects with R/R HNSCC who have disease progression after receiving at least 1 platinum-based chemotherapy and at least 1 anti-programmed death receptor protein-1 (PD-1)/anti-programmed death-ligand 1 (PD-L1) therapy, whether in combination or separately. In Part 2, subjects will be randomized in a ratio of 2:1 to receive either GSK3359609 in combination with tremelimumab at the recommended Phase 2 dose or investigators choice of a single-agent standard of care (SOC) therapy including paclitaxel, docetaxel or cetuximab. The total duration of subjects in the study will be approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.
* Male or female, aged 18 years or older.
* Body weight >=30 kilograms (kg).
* Histological or cytological documentation of an invasive malignancy that was diagnosed as locally advanced/metastatic or relapsed/refractory and is of one of the following tumor types: a) Part 1: cutaneous melanoma; HNSCC (oral cavity, larynx, oropharynx, hypopharynx, nasal cavity/paranasal sinuses); non-small cell lung cancer (squamous and non-squamous); urothelial carcinoma of the upper and lower urinary tract; clear cell renal carcinoma; castrate resistant prostate adenocarcinoma. b) Part 2: HNSCC (oral cavity, larynx, pharynx, paranasal sinuses).
* Part 1 only: Disease that has progressed after standard therapy for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate, or if no further standard therapy exists, or where standard therapy is refused. May be anti-PD-1/anti-PD-L1 experienced or naïve.
* Part 2 only: Disease that has progressed after receiving platinum-based chemotherapy (unless medically contraindicated or discontinued due to toxicity) and anti-PD-1/anti-PD-L1 therapy (in combination or as separate lines of therapy in either sequence).
* Measurable disease per RECIST version 1.1 guidelines. Palpable lesions that are not measurable by radiographic or photographic evaluations may not be utilized as the only measurable lesion. Any measurable lesion biopsied at Screening cannot be followed as a target/index lesion unless agreed upon by GlaxoSmithKline (GSK).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* Adequate organ function.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions apply: a) Not a woman of childbearing potential (WOCBP); or, b) A WOCBP who agrees to follow the contraceptive while receiving study intervention and for at least 180 days after the last dose of study intervention.
* A male subject must agree to use a highly effective contraception while receiving study intervention and for at least 180 days after the last dose of study intervention and refrain from donating sperm during this period.
* Agree to collection of tumor tissue: a) Part 1 and Part 2: Archival tumor tissue collected any time from the initial diagnosis of invasive malignancy; a fresh tumor biopsy will be required if archival specimen is unavailable prior to first dose. b) Part 1 pharmacokinetic/pharmacodynamic cohort(s): Archival tissue as noted in point (a) above. Paired tumor biopsies: tumor tissue collected any time after completion of dosing of the last therapy and prior to first dose and an on-treatment biopsy. c) Part 2: A minimum of 15 subjects from each arm will be required to provide paired tumor biopsies (in addition to the archival tissues as noted in point (a) above): tumor tissue collected any time after completion of dosing of the last therapy and prior to first dose and an on-treatment biopsy.

Exclusion Criteria:

* Received prior treatment with the following therapies; calculation is based on date of last therapy to date of first dose of study intervention or SOC: a) Cytotoxic T-Lymphocyte-Associated Protein 4 (CTLA-4 [including tremelimumab] or Inducible T Cell Co-Stimulator (ICOS)-directed therapies at any time; b) >=4 lines of prior anticancer treatment: In subjects that relapse or progress within 1 year from the beginning of adjuvant or concurrent therapy, the adjuvant/concurrent therapy is considered first line therapy; c) Systemic anticancer therapy or investigational therapy within 30 days, or 5 half-lives, whichever is shorter; at least 14 days must have elapsed between the date of the last prior therapy to the date of first dose of study intervention or SOC.
* Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment per RECIST v1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. At least 14 days must have elapsed between the date of the last dosage of radiation and the first dose of study intervention/SOC.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last two years, except: a) Any other invasive malignancy for which the subject was definitively treated, has been disease-free for <=2 years and in the opinion of the Investigator and Medical Monitor will not affect the evaluation of the effects of the study intervention or SOC on the currently targeted malignancy, may be included in this clinical study; Curatively treated non-melanoma skin cancer or successfully treated in-situ carcinoma.
* Toxicity from previous anticancer treatment that includes: a) >=Grade 3 toxicity considered related to prior immunotherapy and that led to treatment discontinuation; b) Toxicity related to prior treatment that has not resolved to <=Grade 1 (except alopecia, vitiligo, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <=Grade 2).
* Central nervous system (CNS) metastases, with the following exception: Subjects with previously treated CNS metastases who are clinically stable and had no requirement for steroids during at least 14 days prior to first dose of study intervention or SOC.
* Major surgery <=28 days of first dose of study intervention or SOC.
* Autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years. Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (i.e., adrenal insufficiency) are not considered systemic treatments.
* Recent history (within 24 weeks) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* Receiving systemic steroids (>=10 milligrams [mg] oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to first dose of study intervention or SOC.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* Received live-virus vaccine within 30 days from start of study intervention or SOC.
* Current or history of idiopathic pulmonary fibrosis, pneumonitis (for past, subject is excluded if steroids were required), interstitial lung disease or organizing pneumonia.
* Recent history (within 24 weeks) of uncontrolled, symptomatic ascites, pleural or pericardial effusions.
* History or evidence of cardiac abnormalities within the 24 weeks prior to enrollment which include: a) Serious uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block. b) Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting. c) Symptomatic pericarditis.
* Current unstable liver or biliary disease per Investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy.
* Known human immunodeficiency virus infection; positive test for hepatitis B active infection (presence of hepatitis B surface antigen) or hepatitis C active infection.
* History of severe hypersensitivity to monoclonal antibodies, the Standard of Care agents, including any ingredient used in the formulation, based on which treatment the subject is to receive.
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
* For subjects receiving SOC: Requires therapy with a medication that may alter the PK of the SOC agent (e.g., strong inducers or inhibitors of cytochrome P (CYP)3A4 for subjects receiving docetaxel or paclitaxel) during the study treatment period. Please refer to the package insert for the agent the subject is to receive.
* For subjects receiving SOC: Any contraindication, per the package insert and/or Institutional guidelines, to the treatment the subject is to receive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Hilton JF, Ott PA, Hansen AR, Li Z, Mathew M, Messina CH, Dave V, Ji X, Karpinich NO, Hirschfeld S, Ballas M, Zandberg DP. INDUCE-2: A Phase I/II, open-label, two-part study of feladilimab in combination with tremelimumab in patients with advanced solid tumors. Cancer Immunol Immunother. 2024 Feb 13;73(3):44. doi: 10.1007/s00262-023-03623-z. PMID 38349570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States and Canada.
Pre-assignment Details: The results presented are for Part 1 of the study. Part 2 was not initiated due to Sponsor decision to not proceed based on scientific and portfolio priority reasons and lack of adequate efficacy and not due to safety reasons in Part 1. A total of 26 participants were enrolled in this study.
Groups:
- Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 8 milligram (mg) Feladilimab first as a 30-minute intravenous (IV) infusion once every 3 weeks (Q3W) in combination with 75 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once every 12 weeks (Q12W).
- Part 1: Feladilimab 24 mg + Tremelimumab 75 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 24 mg Feladilimab first as a 30-minute IV infusion once Q3W in combination with 75 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once Q12W.
- Part 1: Feladilimab 8 mg + Tremelimumab 225 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 8 mg Feladilimab first as a 30-minute IV infusion once Q3W in combination with 225 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once Q12W.
- Part 1: Feladilimab 80 mg + Tremelimumab 75 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 80 mg Feladilimab first as a 30-minute IV infusion once Q3W in combination with 75 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once Q12W.
- Part 1: Feladilimab 24 mg + Tremelimumab 225 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 24 mg Feladilimab first as a 30-minute IV infusion once Q3W in combination with 225 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once Q12W.
- Part 2: Feladilimab +Tremelimumab: In Part 2, participants with Head and Neck Squamous Cell Carcinoma (HNSCC) who have progressed after receiving at least 1 platinum-based chemotherapy and at least one anti- Programmed death receptor protein-1 (PD-1)/ Programmed death-ligand 1 (PD-L1) therapy, whether in combination or separately were planned to be enrolled. Participants were planned to be administered with Feladilimab and Tremelimumab as an IV infusion after the Recommended Phase 2 Dose (RP2D) determination.
- Part 2: Standard of Care (SOC): In Part 2, participants with HNSCC who have progressed after receiving at least 1 platinum-based chemotherapy and at least one anti-PD-1/PD-L1 therapy, whether in combination or separately were planned to be enrolled. Participants were planned to be administered a single agent SOC therapy of either paclitaxel (as an IV infusion once weekly at a dose of 80 milligrams per meter square (mg/m^2)), docetaxel (as an IV infusion once Q3W at a dose of 75 mg/m^2) or cetuximab (at a loading dose of 400 mg/m^2 followed by 250 mg/m^2 once weekly) as per the investigator's choice.
Period: Overall Study
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg | Part 2: Feladilimab +Tremelimumab | Part 2: Standard of Care (SOC)
Started | 1 | 1 | 5 | 3 | 16 | 0 | 0
Completed | 1 | 0 | 4 | 3 | 10 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Groups:
- Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg: In Part 1, participants with advanced, selected solid tumors were enrolled. Participants were administered 8 mg Feladilimab first as a 30-minute IV infusion once Q3W in combination with 75 mg tremelimumab as an IV infusion over 60 minutes beginning at least 1 hour and no more than 2 hours once Q3W for 6 doses followed by once Q12W.
- Part 2: Feladilimab + Tremelimumab: In Part 2, participants with HNSCC who have progressed after receiving at least 1 platinum-based chemotherapy and at least one anti-PD-1/ PD-L1 therapy, whether in combination or separately were planned to be enrolled. Participants were planned to be administered with Feladilimab and Tremelimumab as an IV infusion after the RP2D determination.
- Part 2: Standard of Care (SOC): In Part 2, participants with HNSCC who have progressed after receiving at least 1 platinum-based chemotherapy and at least one anti-PD-1/PD-L1 therapy, whether in combination or separately were planned to be enrolled. Participants were planned to be administered with a single agent SOC therapy of either paclitaxel (as an IV infusion once weekly at a dose of 80 mg/m^2), docetaxel (as an IV infusion once every 3 weeks at a dose of 75 mg/m^2) or cetuximab (at a loading dose of 400 mg/m^2 followed by 250 mg/m^2 once weekly) as per the investigator's choice.
- Total: Total of all reporting groups
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC) | Total
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16 | 0 | 0 | 26
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 51.0 (0) | 51.0 (0) | 58.2 (11.73) | 69.0 (12.77) | 66.8 (11.51) |  |  | 64.2 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 0 | 4 | 0 | 0 | 9
  Male | 0 | 0 | 2 | 3 | 12 | 0 | 0 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Multiple | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 1 | 1 | 5 | 3 | 14 | 0 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)-Part 1
Description: A DLT is considered by the investigator to be clinically relevant, attributed event within first 28 days of intervention meeting the following criteria of toxicity, Hematologic: Febrile neutropenia, Grade 4 neutropenia of greater than (>) 7 days in duration or requiring Granulocyte- Colony stimulating factor (G-CSF), Grade 4 anemia and Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia; Non-hematologic: Grade 4 toxicity, Grade 3 pneumonitis, any greater than or equal to (≥) Grade 2 pneumonitis that does not resolve to less than or equal to (≤ ) Grade 1 within 3 days of the initiation of maximal supportive care, Grade 3 toxicity that does not resolve to Grade 1 or baseline within 3 days despite optimal supportive care and any Grade 2 ocular toxicity requiring systemic steroids, or any ≥ Grade 3 ocular toxicity.
Time Frame: Up to 28 days
Population: All Treated Population includes all participants who received at least 1 dose of Tremelimumab or Feladilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With DLTs According to Severity-Part 1
Description: The severity of all toxicities were graded using the National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 5.0. Grade 1: Mild reaction; infusion interruption not indicated; intervention not indicated; Grade 2: Requires therapy or infusion interruption but responds promptly to symptomatic treatment or prophylactic medications indicated for ≤24 hours; Grade 3: Prolonged (i.e., not rapidly responsive to symptomatic medication and/or brief interruption of infusion) or recurrence of symptoms following initial improvement; hospitalization indicated for other clinical sequelae; Grade 4: Life-threatening; pressor or ventilatory support indicated; Grade 5: Death related to AE.
Time Frame: Up to 28 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)-Part 1
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect and important medical events may jeopardize the subject or may require medical or surgical intervention/SOC to prevent one of the other outcomes mentioned before. AESIs are defined as events of potential immunologic etiology, including immune related AEs.
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  AEs | 1 | 1 | 5 | 3 | 16
  SAEs | 0 | 0 | 3 | 3 | 6
  AESIs | 0 | 0 | 2 | 0 | 7

4. Primary Outcome: Number of Participant With AE/SAE/DLTs Leading to Dose Modifications/Delays/Withdrawals-Part 1
Description: The number of participants with AE/SAE/DLTs leading to dose modifications/delays/withdrawals were summarized.
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Any Aes-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any Aes-Dose Delay | 0 | 0 | 3 | 0 | 4
  Any Aes-Dose Withdrawal | 0 | 0 | 1 | 0 | 3
  Any SAEs-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any SAEs-Dose Delay | 0 | 0 | 1 | 0 | 1
  Any SAEs-Dose Withdrawal | 0 | 0 | 1 | 0 | 2
  Any DLTs-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any DLTs-Dose Delay | 0 | 0 | 0 | 0 | 1
  Any DLTs-Dose Withdrawal | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With AEs, SAEs, AESIs According to Severity - Part 1
Description: as for outcome 2
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Grade 1: AEs | 0 | 0 | 0 | 0 | 4
  Grade 2: AEs | 1 | 1 | 1 | 0 | 4
  Grade 3: AEs | 0 | 0 | 3 | 3 | 6
  Grade 4: AEs | 0 | 0 | 1 | 0 | 1
  Grade 5: AEs | 0 | 0 | 0 | 0 | 1
  Grade 1: SAEs | 0 | 0 | 0 | 0 | 0
  Grade 2: SAEs | 0 | 0 | 0 | 0 | 1
  Grade 3: SAEs | 0 | 0 | 2 | 3 | 3
  Grade 4: SAEs | 0 | 0 | 1 | 0 | 1
  Grade 5: SAEs | 0 | 0 | 0 | 0 | 1
  Grade 1: AESI | 0 | 0 | 0 | 0 | 3
  Grade 2: AESI | 0 | 0 | 2 | 0 | 2
  Grade 3: AESI | 0 | 0 | 0 | 0 | 1
  Grade 4: AESI | 0 | 0 | 0 | 0 | 1
  Grade 5: AESI | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Severe- AEs/SAEs/DLTs Leading to Dose Modifications/Delays/Withdrawals-Part 1
Description: The number of participants with severe- AE/SAE/DLTs leading to dose modifications/delays/withdrawals were summarized.
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Any Severe Aes-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any Severe Aes-Dose Delay | 0 | 0 | 3 | 0 | 4
  Any Severe Aes-Dose Withdrawal | 0 | 0 | 1 | 0 | 3
  Any Severe SAEs-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any Severe SAEs-Dose Delay | 0 | 0 | 1 | 0 | 1
  Any Severe SAEs-Dose Withdrawal | 0 | 0 | 1 | 0 | 2
  Any Severe DLTs-Dose Modification | 0 | 0 | 0 | 0 | 0
  Any Severe DLTs-Dose Delay | 0 | 0 | 0 | 0 | 1
  Any Severe DLTs-Dose Withdrawal | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)-Part 1
Description: SBP and DBP were measured after 5 minutes of rest for the participant.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Millimeters of mercury (mmHg)
  SBP, Baseline (Day 1) | 104 | 128 | 128 (14.967) | 133.67 (11.676) | 127.5 (16.415)
  SBP, Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  SBP, Week 4 | 16 | -12 | -10 (11.726) | -12 (11.533) | -0.27 (19.568)
  DBP, Baseline (Day 1) | 73 | 79 | 83.4 (8.081) | 74.67 (4.041) | 76.25 (9.015)
  DBP, Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  DBP, Week 4 | 4 | -3 | -5 (3.162) | -4 (6.557) | -2.8 (7.552)

8. Primary Outcome: Change From Baseline in Temperature-Part 1
Description: Temperature was measured after 5 minutes of rest for the participant.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Celsius (C)
  Baseline (Day 1) | 36.5 | 36.9 | 36.8 (0.212) | 36.6 (0.173) | 36.64 (0.479)
  Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Week 4 | 0 | -0.3 | 0.04 (0.321) | 0.2 (0.1) | 0.04 (0.378)

9. Primary Outcome: Change From Baseline in Pulse Rate-Part 1
Description: Pulse rate was measured after 5 minutes of rest for the participant.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
beats/minute
  Baseline (Day 1) | 81 | 83 | 91.6 (29.771) | 79.67 (9.074) | 76.56 (14.724)
  Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Week 4 | 1 | 0 | -2.4 (20.732) | 5 (15.716) | 8.07 (10.747)

10. Primary Outcome: Change From Baseline in Respiratory Rate-Part 1
Description: Respiratory rate was measured after 5 minutes of rest for the participant.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: breaths/ minute
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
breaths/ minute
  Baseline (Day 1) | 18 | 18 | 17.6 (0.894) | 16 (0) | 16.75 (1.065)
  Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Week 4 | 0 | -2 | 0 (1.414) | 2 (0) | 0.07 (1.668)

11. Primary Outcome: Change From Baseline in Oxygen Saturation-Part 1
Description: Oxygen saturation was measured using pulse oximeter after 5 minutes of rest for the participant.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage (%) of Oxygen
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Percentage (%) of Oxygen
  Baseline (Day 1) | 96 | 95 | 95.6 (2.881) | 96 (1.00) | 97.63 (1.586)
  Week 4: number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Week 4 | 2 | 5 | 0.8 (1.304) | 0 (2.00) | -0.2 (2.007)

12. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: Single 12-lead ECG was obtained using an automated ECG machine. ECG findings were categorized as: normal, abnormal - clinically significant (CS), or abnormal - not clinically significant (NCS), as determined by the investigator.
Time Frame: Baseline (Pre dose, Day 1) and up to 4 Years
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Baseline (Pre dose, Day 1): Normal | 1 | 1 | 1 | 1 | 6
  Baseline (Pre dose, Day 1): Abnormal CS | 0 | 0 | 1 | 0 | 0
  Baseline (Pre dose, Day 1): Abnormal NCS | 0 | 0 | 3 | 2 | 10
  Worst case Post-Baseline: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  Worst case Post-Baseline: Normal | 0 | 0 | 0 | 1 | 0
  Worst case Post-Baseline: Abnormal CS | 0 | 0 | 0 | 0 | 0
  Worst case Post-Baseline: Abnormal NCS | 0 | 0 | 0 | 1 | 2

13. Primary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil and Platelet Count-Part 1
Description: Blood samples were collected to assess change from Baseline in neutrophil, lymphocyte, monocyte, eosinophil, basophil and platelet counts.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
10^9 cells/liter
  Basophils, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 4 | 2 | 13
  Basophils, Baseline (Day 1) | 0.00 | 0.00 | 0.05 (0.0577) | 0.01 (0.0141) | 0.039 (0.048)
  Basophils, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 2 | 10
  Basophils, Week 4 | 0.00 |  | 0 (0) | 0.005 (0.0071) | 0.007 (0.0344)
  Eosinophils, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 4 | 2 | 13
  Eosinophils, Baseline (Day 1) | 0.3 | 0.1 | 0.35 (0.173) | 0.08 (0.113) | 0.2 (0.217)
  Eosinophils, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 2 | 10
  Eosinophils, Week 4 | 0.4 |  | 0.03 (0.15) | 0.06 (0.064) | 0.07 (0.169)
  Lymphocytes, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 4 | 2 | 13
  Lymphocytes, Baseline (Day 1) | 1 | 1.5 | 0.9 (0.216) | 1.25 (0.212) | 0.92 (0.223)
  Lymphocytes, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 2 | 9
  Lymphocytes, Week 4 | 0.4 |  | 0.23 (0.15) | -0.38 (0.46) | 0.01 (0.185)
  Monocytes, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 4 | 2 | 13
  Monocytes, Baseline (Day 1) | 0.4 | 0.3 | 0.8 (0.2944) | 1.255 (0.9122) | 0.738 (0.3004)
  Monocytes, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 2 | 10
  Monocytes, Week 4 | 0 |  | 0.05 (0.1732) | -0.215 (0.1202) | 0.038 (0.2598)
  Neutrophils, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 4 | 2 | 13
  Neutrophils, Baseline (Day 1) | 4 | 3.9 | 4.38 (1.548) | 6.2 (2.97) | 11.32 (21.379)
  Neutrophils, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 2 | 9
  Neutrophils, Week 4 | 0.3 |  | 0.93 (0.512) | -0.9 (0.7) | -8.95 (26.151)
  Platelets, Baseline (Day 1) | 196 | 325 | 250.6 (103.5) | 229.7 (147.06) | 266.3 (90.28)
  Platelets, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Platelets, Week 4 | -1 |  | 8.6 (34.93) | -8.7 (16.65) | 31.3 (42.72)

14. Primary Outcome: Change From Baseline in Hemoglobin Level-Part 1
Description: Blood samples were collected to assess change from baseline in hemoglobin level.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
grams/liter
  Baseline (Day 1) | 125 | 134 | 123.4 (32.61) | 125 (23.07) | 111.5 (12.74)
  Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Week 4 | 5 |  | -5.8 (4.21) | 0.3 (2.89) | -0.7 (10.78)

15. Primary Outcome: Change From Baseline in Hematocrit Level-Part 1
Description: Blood samples were collected to assess change from baseline in hematocrit level.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: fraction of 1
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
fraction of 1
  Baseline (Day 1) | 0.38 | 0.4 | 0.385 (0.10999) | 0.3937 (0.0647) | 0.3421 (0.03603)
  Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Week 4 | 0 |  | -0.0202 (0.01494) | -0.0017 (0.01102) | -0.0039 (0.03413)

16. Primary Outcome: Change From Baseline in Erythrocytes Count-Part 1
Description: Blood samples were collected to assess change from baseline in Erythrocytes count.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
10^12 cells/liter
  Baseline (Day 1) | 4.2 | 4.65 | 4.328 (1.2592) | 4.673 (0.4885) | 3.76 (0.526)
  Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Week 4 | 0.13 |  | -0.216 (0.2131) | 0.04 (0.1652) | 0.016 (0.3913)

17. Primary Outcome: Change From Baseline in Albumin and Total Protein Levels-Part 1
Description: Blood samples were collected to assess change from Baseline in albumin and total protein levels.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: grams/Liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
grams/Liter
  Albumin, Baseline (Day 1) | 41 | 40 | 36 (7.18) | 36.7 (9.24) | 37.9 (2.79)
  Albumin, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Albumin, Week 4 | 0 |  | 0 (3.81) | -0.7 (2.31) | -2.1 (2.81)
  Protein, Baseline (Day 1): number analyzed (Participants) | 1 | 0 | 3 | 3 | 16
  Protein, Baseline (Day 1) | 71 |  | 66.7 (7.02) | 73 (3.61) | 72.1 (6.51)
  Protein, Week 4: number analyzed (Participants) | 0 | 0 | 3 | 3 | 13
  Protein, Week 4 |  |  | 3.3 (2.89) | 0 (4.36) | 1.4 (4.31)

18. Primary Outcome: Change From Baseline in Creatinine and Bilirubin Levels-Part 1
Description: Blood samples were collected to assess change from baseline in creatinine and bilirubin levels.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles/ Liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
micromoles/ Liter
  Bilirubin, Baseline (Day 1) | 5 | 7 | 6.1 (2.44) | 6.1 (2.84) | 6.5 (4.23)
  Bilirubin, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Bilirubin, Week 4 | -1 |  | 2.2 (2.48) | -1.1 (1.97) | -0.4 (1.52)
  Creatinine, Baseline (Day 1) | 59000 | 63000 | 31636.7 (43702.44) | 73.5 (33.52) | 93 (44.72)
  Creatinine, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Creatinine, Week 4 | 1000 |  | -1798.9 (3493.56) | 3.1 (4.29) | -2.9 (9.53)

19. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), Lactate Dehydrogenase (LDH) Levels-Part 1
Description: Blood samples were collected to assess change from baseline in ALT, AST ALP, LDH levels.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units/milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
International Units/milliliter
  ALP, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 5 | 2 | 13
  ALP, Baseline (Day 1) | 53 | 68 | 307.4 (416.93) | 121.5 (82.73) | 120.2 (60.54)
  ALP, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 2 | 11
  ALP, Week 4 | 2 |  | 55.8 (101.74) | -18 (25.46) | 36.2 (75.58)
  ALT, Baseline (Day 1) | 18 | 25 | 24 (14.18) | 26.7 (24.79) | 18.2 (13.49)
  ALT, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  ALT, Week 4 | -2 |  | 8.2 (13.05) | -4.7 (15.14) | 7.4 (26.46)
  AST, Baseline (Day 1) | 32 | 44 | 24.6 (9.91) | 23.7 (15.89) | 21.9 (8.23)
  AST, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  AST, Week 4 | 0 |  | 10 (14.2) | -7 (14.73) | 12.9 (35.1)
  LDH, Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  LDH, Baseline (Day 1) | 325 | 382 | 228.8 (20.69) | 168 (104.23) | 239.9 (139.36)
  LDH, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 10
  LDH, Week 4 | 127 |  | 11.4 (42.76) | 31.3 (53.3) | 42.9 (85.66)

20. Primary Outcome: Change From Baseline in Amylase and Lipase Levels-Part 1
Description: Blood samples were collected to assess change from baseline in amylase and lipase levels.
Time Frame: Baseline (Day 1) and week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units/milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Units/milliliter
  Amylase, Baseline (Day 1) | 48 | 50 | 50.2 (34.85) | 40 (15.62) | 51.5 (26.72)
  Amylase, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 3 | 15
  Amylase, Week 4 | -2 |  | -5.3 (7.23) | -5 (1) | -3.5 (9.64)
  Lipase, Baseline (Day 1) | 28 | 23 | 50.8 (55.65) | 54.7 (48.99) | 34.6 (27.8)
  Lipase, Week 4: number analyzed (Participants) | 1 | 0 | 4 | 3 | 15
  Lipase, Week 4 | 0 |  | 1.5 (4.65) | -13 (23.81) | 6.1 (35.96)

21. Primary Outcome: Change From Baseline in Urea, Glucose, Potassium, Sodium and Calcium Levels-Part 1
Description: Blood samples were collected to assess change in levels of urea, glucose, potassium, sodium and calcium from baseline.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles/Liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
millimoles/Liter
  Glucose, Baseline (Day 1) | 6.7 | 7.3 | 6.09 (1.6994) | 5.897 (0.2754) | 6.397 (1.5963)
  Glucose, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Glucose, Week 4 | -0.3 |  | -0.365 (1.3225) | -0.848 (0.4949) | -0.11 (1.0164)
  Calcium, Baseline (Day 1) | 2.37 | 2.24 | 2.325 (0.1221) | 2.397 (0.1475) | 2.33 (0.0886)
  Calcium, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Calcium, Week 4 | 0.15 |  | 0.137 (0.1385) | 0.05 (0.1322) | -0.028 (0.0878)
  Potassium, Baseline (Day 1) | 4.3 | 4 | 4.18 (0.606) | 4.3 (0.173) | 4.22 (0.391)
  Potassium, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Potassium, Week 4 | -0.3 |  | 0.04 (0.586) | -0.03 (0.306) | -0.01 (0.328)
  Sodium, Baseline (Day 1) | 138 | 140 | 137.2 (4.49) | 137.3 (3.21) | 137.1 (3.52)
  Sodium, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Sodium, Week 4 | -1 |  | 0.2 (1.3) | 0.7 (0.58) | -1 (2.65)
  Urea, Baseline (Day 1) | 3.4 | 3.3 | 6.36 (1.226) | 7.36 (0.75) | 6.92 (3.495)
  Urea, Week 4: number analyzed (Participants) | 1 | 0 | 5 | 3 | 13
  Urea, Week 4 | 1.5 |  | -1.37 (1.09) | 1.08 (0.357) | -0.51 (1.633)

22. Primary Outcome: Change From Baseline in Specific Gravity of Urine-Part 1
Description: Urine samples were collected to assess change from baseline in specific gravity of urine.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Ratio
  Baseline (Day 1) | 1.015 | 1.02 | 1.0204 (0.00856) | 1.021 (0.01015) | 1.0159 (0.00605)
  Week 4: number analyzed (Participants) | 1 | 0 | 4 | 3 | 15
  Week 4 | 0.005 |  | -0.0055 (0.00666) | 0.0013 (0.00115) | -0.0005 (0.006)

23. Primary Outcome: Change From Baseline in Potential of Hydrogen (pH) of Urine-Part 1
Description: Urine samples were collected to assess change from baseline in pH of urine.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
pH
  Baseline (Day 1) | 6.5 | 7 | 6 (1.173) | 5.33 (0.289) | 6.16 (0.826)
  Week 4: number analyzed (Participants) | 1 | 0 | 4 | 3 | 15
  Week 4 | -0.5 |  | 0.5 (0.707) | -0.33 (0.289) | -0.24 (0.918)

24. Primary Outcome: Number of Participants With Abnormal Urinalysis Parameters-Part 1
Description: The dipstick test gives positive or negative results for protein, ketones, occult blood and glucose in urine. Positive test results were considered as abnormal. Number of participants with positive test results have been summarized.
Time Frame: Week 4
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 0 | 5 | 3 | 16
Participants
  Dip stick test for Glucose | 0 |  | 1 | 0 | 2
  Dip stick test for Protein | 0 |  | 1 | 0 | 6
  Dip stick test for Occult Blood | 1 |  | 2 | 1 | 5
  Dip stick test for Ketones | 0 |  | 4 | 0 | 3

25. Primary Outcome: Change From Baseline in Thyroid Stimulating Hormone (TSH) or Thyrotropin-Part 1
Description: Blood samples were collected to assess change from Baseline in TSH.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: milliUnits/Liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
milliUnits/Liter
  Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Baseline (Day 1) | 0.79 | 1.22 | 1.856 (1.6061) | 1.463 (1.2079) | 2.211 (1.7527)
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 4 |  |  |  | -0.87 |

26. Primary Outcome: Change From Baseline in Free Triiodothyronine (T3)-Part 1
Description: Blood samples were collected to assess change from Baseline in free T3.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Picomoles per liter
  Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 2 | 1 | 9
  Baseline (Day 1) | 3.5 | 3.6 | 2.75 (0.212) | 4.47 | 3.88 (0.665)
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Change From Baseline in Free Thyroxine (T4)-Part 1
Description: Blood samples were collected to assess change from baseline in free T4.
Time Frame: Baseline (Day 1) and Week 4
Population: All Treated Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Picomoles per liter
  Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 5 | 3 | 15
  Baseline (Day 1) | 10 | 11 | 12.43 (3.128) | 13.84 (2.296) | 15.98 (3.144)
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 4 |  |  |  | 2.57 |

28. Primary Outcome: Overall Survival-Part 2
Description: For participants in Part 2, overall survival is defined as time from the date of randomization to the date of death due to any cause.
Time Frame: Up to 4 years
Population: Intent-To-Treat population includes all participants in Part 2 who were planned to be randomized in the trial. Part 1 participants that were dosed at the dose level chosen for expansion in Part 2 were planned to be excluded from the Part 2 ITT. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Overall Response Rate-Part 1
Description: Overall response rate is defined as percentage of participants with confirmed complete response (Disappearance of all target lesions. Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 millimeter [mm]) or partial response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) at any time as per response evaluation criteria in solid tumors (RECIST) version 1.1.
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Percentage of Participants | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 52.2] | 0 [0 to 70.8] | 6.3 [0.2 to 30.2]

30. Secondary Outcome: Overall Response Rate-Part 2
Description: Overall response rate is defined as percentage of participants with confirmed complete response (Disappearance of all target lesions. Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm) or partial response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) at any time as per RECIST version 1.1.
Time Frame: Up to 4 years
Population: Intent-To-Treat Population. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Disease Control Rate-Part 1
Description: Disease control rate is defined as percentage of subjects with confirmed complete response (Disappearance of all target lesions. Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm) or partial response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) or at least 18 weeks of stable disease (Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) as per RECIST version 1.1.
Time Frame: Up to 4 years
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Percentage of Participants | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 52.2] | 33.3 [0.8 to 90.6] | 12.5 [1.6 to 38.3]

32. Secondary Outcome: Disease Control Rate-Part 2
Description: as for outcome 31
Time Frame: Up to 4 years
Population: as for outcome 30
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Progression Free Survival-Part 2
Description: For Part 2, progression free survival duration is defined as the time from the date of randomization to first documented evidence of disease progression (At least a 20% increase in the sum of diameters of target lesions and In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm) or death (regardless of cause of death), whichever comes first as per RECIST version 1.1.
Time Frame: Up to 4 years
Population: as for outcome 30
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Time to Response-Part 2
Description: Time to response is defined as the time from the first dose to the first documented evidence of complete response (Disappearance of all target lesions. Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm) or partial response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) for participants with a confirmed CR or PR as per RECIST version 1.1.
Time Frame: Up to 4 years
Population: as for outcome 30
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Duration of Response-Part 2
Description: Duration of response is defined as time from the first documented evidence of response until the first documented sign of disease progression or death among participants who achieve a response (CR [Disappearance of all target lesions. Any pathological lymph nodes {whether target or non-target} must have reduction in short axis to <10 mm or PR [At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters] as per RECIST version 1.1).
Time Frame: Up to 4 years
Population: as for outcome 30
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Feladilimab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic (PK) Population includes all participants from the All Treated population for whom at least one PK sample was obtained, analysed and measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
nanograms/milliliter | 2758 | 5965 | 2686.6 (25.7) | 28340.9 (12.3) | 6098.3 (25.3)

37. Secondary Outcome: Cmax of Tremelimumab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 0 | 16
nanograms/milliliter | 0 | 0 | 112312.1 (8.2) |  | 93206.7 (24.8)

38. Secondary Outcome: Cmax of Feladilimab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose at Weeks 1, 2, 4, 7, 10, 13, 16, 19, 25, then every 12 weeks for 2 years; end of infusion at Weeks 1, 19 and 25; and 4 hours post-infusion at Week 1
Population: Pharmacokinetic Population. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Cmax of Tremelimumab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment.
Time Frame: as for outcome 38
Population: as for outcome 38
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Feladilimab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/ milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 0 | 5 | 3 | 16
nanograms/ milliliter | 462 |  | 348 (14.2) | 3197 (31) | 856.4 (35.9)

41. Secondary Outcome: Cmin of Tremelimumab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/ milliliter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 0 | 5 | 3 | 16
nanograms/ milliliter | 6467 |  | 22466.3 (58.4) | 5715.6 (43.9) | 15084.9 (48.4)

42. Secondary Outcome: Cmin of Feladilimab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose at Weeks 1, 2, 4, 7, 10, 13, 16, then every 12 weeks for 2 years; end of infusion; and 4 hours post-infusion at Week 1
Population: as for outcome 38
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Cmin of Tremelimumab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment.
Time Frame: as for outcome 42
Population: as for outcome 38
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC[0-t]) of Feladilimab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliLiter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 0 | 5 | 3 | 16
nanograms*hours/milliLiter | 545097.4 |  | 453561.5 (11.7) | 4552653.1 (18.5) | 1055659.5 (23.5)

45. Secondary Outcome: AUC(0-t) of Tremelimumab-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose, end of infusion and 4 hours post dose at Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliLiter
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 9
nanograms*hours/milliLiter |  |  |  |  | 18160725.7 (23.4)

46. Secondary Outcome: AUC(0-t) of Feladilimab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment.
Time Frame: Pre-dose at Weeks 1, 2, 4, 7, 10, 13, 16, 19, 25, then every 12 weeks for 2 years; end of infusion at Weeks 1, 19 and 25, and 4 hours post-infusion at Week 1
Population: as for outcome 38
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: AUC(0-t) of Tremelimumab-Part 2
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic assessment
Time Frame: as for outcome 42
Population: as for outcome 38
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Number of Participants With Anti-drug Antibodies Against Feladilimab-Part 1
Description: Serum samples were collected and tested for the presence of antibodies to feladilimab.
Time Frame: Pre-dose at Week 4, 7, 10 and 13
Population: All Treated population. Only those participants with data available at specified time points has been analyzed. Number of participants analyzed refers to the analysis population. Number analyzed at each time point refers to the participants for whom screening assays were conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Week 4: number analyzed (Participants) | 1 | 0 | 3 | 3 | 15
  Week 4 | 0 | 0 | 1 | 0 | 5
  Week 7: number analyzed (Participants) | 1 | 1 | 3 | 3 | 12
  Week 7 | 0 | 0 | 1 | 0 | 2
  Week 10: number analyzed (Participants) | 1 | 1 | 3 | 1 | 8
  Week 10 | 0 | 0 | 1 | 0 | 1
  Week 13: number analyzed (Participants) | 1 | 0 | 2 | 2 | 4
  Week 13 | 0 | 0 | 0 | 0 | 1

49. Secondary Outcome: Number of Participants With Anti-drug Antibodies Against Tremelimumab-Part 1
Description: Serum samples were collected and tested for the presence of antibodies to tremelimumab.
Time Frame: Pre-dose at Week 1, 4, 7, 10 and 13
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 16
Participants
  Week 1: number analyzed (Participants) | 1 | 1 | 5 | 2 | 15
  Week 1 | 0 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 1 | 0 | 3 | 3 | 15
  Week 4 | 0 | 0 | 0 | 1 | 2
  Week 7: number analyzed (Participants) | 1 | 1 | 3 | 3 | 12
  Week 7 | 0 | 1 | 0 | 0 | 1
  Week 10: number analyzed (Participants) | 1 | 1 | 3 | 1 | 8
  Week 10 | 0 | 1 | 0 | 0 | 0
  Week 13: number analyzed (Participants) | 1 | 0 | 2 | 2 | 4
  Week 13 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Number of Participants With Anti-drug Antibodies Against Feladilimab-Part 2
Description: Serum samples will be collected and tested for the presence of antibodies to feladilimab.
Time Frame: Up to 2.5 years
Population: ITT Population. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Change From Baseline in Free T4-Part 2
Description: Blood samples will be collected to assess change from baseline in free T4.
Time Frame: Baseline and up to 2 years
Population: All Treated Population. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled.
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Number of Participants With Anti-drug Antibodies Against Tremelimumab-Part 2
Description: Serum samples will be collected and tested for the presence of antibodies to tremelimumab.
Time Frame: Up to 2.5 years
Population: as for outcome 50
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Number of Participants With AEs, SAEs and AESI-Part 2
Description: as for outcome 3
Time Frame: Up to 4 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Number of Participants With AEs, SAEs, AESIs Based on Severity-Part 2
Description: as for outcome 2
Time Frame: Up to 4 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Number of Participants With Severe- AEs/SAEs/DLTs Leading to Dose Modifications/Delays/Withdrawals-Part 2
Description: The number of participants with severe- AE/SAE/DLTs leading to dose modifications/delays/withdrawals were planned to be summarized.
Time Frame: Up to 4 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Change From Baseline in SBP and DBP-Part 2
Description: SBP and DBP will be measured after 5 minutes of rest for the participant.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Change From Baseline in Temperature-Part 2
Description: Temperature will be measured after 5 minutes of rest for the participant.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Change From Baseline in Pulse Rate-Part 2
Description: Pulse rate will be measured after 5 minutes of rest for the participant.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

59. Secondary Outcome: Change From Baseline in Respiratory Rate-Part 2
Description: Respiratory rate will be measured after 5 minutes of rest for the participant.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

60. Secondary Outcome: Change From Baseline in Oxygen Saturation-Part 2
Description: Oxygen saturation will be measured using pulse oximetry after 5 minutes of rest for the participant.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

61. Secondary Outcome: Change From Baseline in ECG Measurement-Part 2
Description: Single 12-lead ECG will be obtained using an automated ECG machine.
Time Frame: Baseline (Pre-dose) up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

62. Secondary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil and Platelet Count-Part 2
Description: Blood samples will be collected to assess change from baseline in neutrophil, lymphocyte, monocyte, eosinophil, basophil and platelet count.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Change From Baseline in Hemoglobin Level-Part 2
Description: Blood samples will be collected to assess change from baseline in hemoglobin level.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Change From Baseline in Hematocrit Level-Part 2
Description: Blood samples will be collected to assess change from baseline in hematocrit level.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Change From Baseline in Erythrocytes Count-Part 2
Description: Blood samples will be collected to assess change from Baseline in erythrocytes count.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

66. Secondary Outcome: Change From Baseline in Albumin and Total Protein Levels-Part 2
Description: Blood samples will be collected to assess change from baseline in albumin and total protein levels.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

67. Secondary Outcome: Change From Baseline in Creatinine and Bilirubin Levels-Part 2
Description: Blood samples will be collected to assess change from baseline in creatinine and bilirubin levels.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

68. Secondary Outcome: Change From Baseline in ALT, AST, ALP, LDH Levels-Part 2
Description: Blood samples will be collected to assess change from baseline in ALT, AST ALP, LDH, amylase and lipase levels.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Change From Baseline in Amylase and Lipase Levels-Part 2
Description: Blood samples were collected to assess change from baseline in amylase and lipase levels.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

70. Secondary Outcome: Change From Baseline in Urea, Glucose, Potassium, Sodium and Calcium Levels -Part 2
Description: Blood samples will be collected to assess change in levels of urea, glucose, potassium, sodium and calcium from baseline.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

71. Secondary Outcome: Change From Baseline in Specific Gravity of Urine-Part 2
Description: Urine samples will be collected to assess change from Baseline in specific gravity of urine.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

72. Secondary Outcome: Change From Baseline in pH of Urine-Part 2
Description: Urine samples will be collected to assess change from baseline in pH of urine.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

73. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters-Part 2
Description: The dipstick test gives positive or negative results for protein, ketones, occult blood and glucose. Positive test results were considered as abnormal. Number of participants with positive test results were planned to be summarized.
Time Frame: Up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

74. Secondary Outcome: Change From Baseline in TSH-Part 2
Description: Blood samples will be collected to assess change from Baseline in TSH.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

75. Secondary Outcome: Change From Baseline in Free T3-Part 2
Description: Blood samples will be collected to assess change from baseline in free T3.
Time Frame: Baseline and up to 2 years
Population: as for outcome 51
Arm/Group | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from Day 1 to upto 4 years
Description: All Treated Population included participants who received at least 1 dose of SOC or tremelimumab or feladilimab. The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled in the same.
Arm/Group | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg | Part 2: Feladilimab + Tremelimumab | Part 2: Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/5 | 0/3 | 1/16 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 3/5 | 3/3 | 6/16 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 5/5 | 3/3 | 16/16 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg (N=1) | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg (N=1) | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg (N=5) | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg (N=3) | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg (N=16) | Part 2: Feladilimab + Tremelimumab (N=0) | Part 2: Standard of Care (SOC) (N=0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Feladilimab (GSK3359609) 8 mg + Tremelimumab 75 mg (N=1) | Part 1: Feladilimab 24 mg + Tremelimumab 75 mg (N=1) | Part 1: Feladilimab 8 mg + Tremelimumab 225 mg (N=5) | Part 1: Feladilimab 80 mg + Tremelimumab 75 mg (N=3) | Part 1: Feladilimab 24 mg + Tremelimumab 225 mg (N=16) | Part 2: Feladilimab + Tremelimumab (N=0) | Part 2: Standard of Care (SOC) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (11) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 10 (10) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor made the decision to not continue the study at the end of Part 1 based on the totality of available data due to lack of efficacy and not due to safety. Hence Part 2 was not initiated and participants were not enrolled in the same.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03693612/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03693612/SAP_001.pdf